CLINICAL TRIAL: NCT05329103
Title: An Early Phase Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of PEEL-224 in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate PEEL-224 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peel Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PEEL-224-001
Record Dates: First submitted 2022-03-31; First posted 2022-04-14 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A: PEEL-224 Dose Escalation (Experimental): PEEL-224 is administered intravenously (IV) on Days 1, 8, and 15 of a 28-day cycle. The study will begin at a low starting dose and will increase between cohorts according to mTPI-2 until a recommended phase 2 dose is determined. Approximately 10 dose levels are anticipated to be studied.
  Interventions: Drug: PEEL-224
- Part 1B: PEEL-224 Dose Confirmation (Experimental): PEEL-224 is administered intravenously (IV) on Days 1 and 15 of a 28-day cycle at the dose determined in Part 1A
  Interventions: Drug: PEEL-224
- Part 2: PEEL-224 plus FOLF+B (Experimental): PEEL-224 is administered intravenously (IV) and in combination with FOLFPB on Days 1 and 15 of a 28-day cycle. Up to 3 dose levels of PEEL-224 will be tested as determined by the results of Part 1.
  Interventions: Drug: PEEL-224; Drug: FOLF+B

INTERVENTIONS:
Drug: PEEL-224 — Lyophilized powder reconstituted with D5W
Drug: FOLF+B — infusional 5-FU, LV, and bevacizumab
  Arms: Part 2: PEEL-224 plus FOLF+B

SUMMARY:
This is a first-in-human, dose escalation, repeat-dose, multi-center, open-label study evaluating safety, tolerability, PK, and preliminary antitumor activity of PEEL-224 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, dose escalation, repeat-dose, multi-center, open-label study evaluating safety, tolerability, PK, and preliminary antitumor activity of a novel topoisomerase I inhibitor (PEEL-224) in patients with advanced solid tumors. Dose escalation will be guided by the modified toxicity probability interval-2 (mTPI-2) design with a target toxicity rate of 25% and an acceptable DLT interval of 20% to 30%. Cohorts of 2 or more patients will be sequentially enrolled at progressively higher dose levels of PEEL-224. For each dose level, all patients must complete Cycle 1 before the decision to dose escalate the next cohort of patients is made.

ELIGIBILITY:
Inclusion criteria:

* Have a diagnosis of colorectal cancer confirmed by local pathology review (histology or cytology) - Part 2 only
* ECOG of 0 or 1
* Have a diagnosis of advanced or metastatic solid tumor that has progressed after prior standard therapy, have been intolerant or ineligible for standard therapy, or have a malignancy for which there is no approved therapy considered standard of care
* Have at least 1 documented measurable lesion as detected by radiological methods at study entry as per Response Evaluation Criteria in Solid Tumors v1.1
* Have adequate bone marrow reserve
* Have adequate liver function
* Have adequate renal function
* Have completed prior anticancer therapy, including investigational agents, ≥28 days or 5 half lives, whichever is shorter, prior to study treatment
* Have resolution of any clinically significant toxic effects of prior therapy

Exclusion criteria:

* Have primary central nervous system tumors
* Have brain or spinal metastases, except if treated by surgery, surgery plus focal radiotherapy, or radiotherapy alone, with no evidence of progression or hemorrhage ≤14 days prior to the first dose of PEEL-224. Have craniospinal radiotherapy ≤12 weeks prior to the first dose of PEEL-224
* Have significant abnormalities in the level of serum electrolytes
* Have received neutrophil growth factor support ≤14 days prior to the first dose of PEEL 224
* Have an active infection ≤14 days prior to the first dose of PEEL-224
* Use of strong cytochrome P450 (CYP)1A2 and CYP3A4 inhibitors and/or inducers ≤14 days prior to the first dose of PEEL-224 or during the study
* Use of systemic corticosteroids ≤14 days prior to the first dose of PEEL-224
* Are known to be HIV-positive, unless CD4 + lymphocyte count ≥ 300/μL, undetectable viral load; AND Receiving anti-retroviral therapy.
* Have uncontrolled hepatitis B infection or hepatitis C infection;
* Are pregnant or lactating, plan to become pregnant, or plan to donate gametes (ova or sperm) for in vitro fertilization during the study period or for 90 days after the patient's last study-related visit (for eligible patients only, if applicable). Eligible female patients unwilling to employ appropriate contraceptive measures to ensure that pregnancy does not occur during the study will be excluded;
* Have evidence of another malignancy ≤2 years prior to screening (except in situ non melanoma skin cell cancers and in situ cervical carcinoma);
* Are currently enrolled in another therapeutic clinical study or a non-therapeutic clinical study that will conflict with scheduled visits required by this study;
* Have clinically significant, uncontrolled cardiovascular disease
* Have history of cerebrovascular accident, transient ischemic attack, or thrombosis requiring treatment ≤3 months prior to the first dose of PEEL-224
* Have received or will receive a live vaccine ≤14 days prior to the first dose of PEEL 224.
* Have tested positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection ≤14 days of the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Determine maximum tolerated dose | 28 days
  Frequency, severity, and relatedness of dose limiting toxicities

SECONDARY OUTCOMES:
Overall safety and tolerability of PEEL-224 | through study completion, expected average of 6 months
  Frequency, severity, and relatedness of AEs and SAEs
Antitumor activity assessment | every 8 weeks through study completion, expected average of 6 months
  based on RECIST 1.1
Cmax of PEEL-224 and its metabolite | Through 96 hours after dosing on Cycle 1 Day 1 and through 168 hours hours of dosing on Cycle 1 Day 15
  maximum blood concentration of PEEL-224 and its metabolite
Tmax of PEEL-224 and its metabolite | Through 96 hours after dosing on Cycle 1 Day 1 and through 168 hours hours of dosing on Cycle 1 Day 15
  Time to maximum blood concentration of PEEL-224 and its metabolite
changes in QTcF/QTcBBB | Through Cycle 1 (28 days)
  ECG parameter readings

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - HonorHealth Research Institiute, Scottsdale, Arizona
  - Stanford Cancer Center, Palo Alto, California
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No